CLINICAL TRIAL: NCT00191425
Title: Comparison of a 2-Year Therapy of Teriparatide Alone and Its Sequential Use for 1 Year, With or Without Raloxifene HCl, in the Treatment of Severe Postmenopausal Osteoporosis
Brief Title: 2-Year Therapy With Teriparatide vs 1-yr Therapy Followed by 1-Year of Raloxifene or Calcium/Vit D in Severe Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6537; B3D-EW-GHCA
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-07-16 (Estimated); Status verified 2007-07

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide; Raloxifene Hydrochloride

INTERVENTIONS:
Drug: Teriparatide
Drug: Raloxifene

SUMMARY:
The primary purpose of the study is to compare 3 different osteoporosis therapies following one year of teriparatide.In the first year,all eligible patients received open-label teriparatide 20 micrograms/day.After 1 year, patients are randomly assigned to one of 3 possible follow-up treatment regimens for the second 12 months: continuation of teriparatide, switch to raloxifene, or no pharmacological treatment(other than the calcium and vitamin D supplements that everyone receives). Patients are stratified into 3 subsets: (a) patients who have never received any anti-osteoporosis treatment before; (b) patients who received prior antiresorptive treatment successfully; (c) patients who failed to respond adequately to prior antiresorptive drugs (such as bisphosphonates or raloxifene) in the past. These latter patients are not randomized at month 12 but will continue treatment with teriparatide 20 micrograms/day throughout the second year.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory women greater or equal to 55 years, at least 2 years postmenopausal.
* Lumbar spine or total hip or femoral neck bone mineral density measurement must be at least 2.5 standard deviations (SD) below the average bone mass for young women (T-score -2.5 or less).
* Presence of at least one known and documented preexisting clinical fragility fracture, in the past 3 years.

Patients may be included in substudy 2 if they meet any one of the following additional criteria - Patients who have sustained at least one new fragility fracture (vertebral or nonvertebral), despite prescription of antiresorptive therapy* during the 12 months prior to the last new fracture or patients who, after a minimum of two years after initiating antiresorptive therapy*, either have a lumbar spine, femoral neck, or total hip BMD of at least - 3SD below the average bone mass for young women (T-score -3 or less), or who show a decrease of at least 3.5% in BMD at any one of these sites.

*Antiresorptive therapy includes all bisphosphonates, raloxifene, ERT/HRT, calcitonin, and vitamin D metabolites.

Exclusion Criteria:

For substudy 1 patients only:

* current or history of vaginal bleeding or spotting of unknown cause in the 1 year prior to study start
* currently suspected or history of venous thrombotic events (VTE), including lower extremity thrombosis, and other major venous thromboses, or high risk of developing VTE as assessment by the investigator.

Treatment with

* Vitamin D >50,000 IU/week or with any dose of calcitriol or vitamin D analogs or agonists in the 6 months prior to visit 2
* Fluorides in the 12 months prior to visit 2.
* Systemic corticosteroids (other than for replacement therapy) in the 1 month prior to visit 2.(Ophthalmic, otic topical, orally inhaled, nasally inhaled, or intra-articular corticosteroid therapy may be used without these restrictions.)

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810
Dates: Start 2002-08; Study Completion 2005-11

PRIMARY OUTCOMES:
Lumbar spine BMD after 24 months.

SECONDARY OUTCOMES:
Hip and femoral neck BMD at 24 months.
Comparison of randomized groups, and descriptive analysis of group receiving open-label treatment with teriparatide for 2 years due to prior antiresorptive treatment failure.
Change in itudinal fracture pattern from 3-year pre-study period to end of the study in all patients who receive teriparatide for 2 years.
Change in back pain after 1, 6, 12, and 24 mths.
Safety of teriparatide.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Pyrmont, Germany

REFERENCES:
- [Derived] Minne H, Audran M, Simoes ME, Obermayer-Pietsch B, Sigurethsson G, Marin F, Dalsky GP, Nickelsen T; EUROFORS Study Group. Bone density after teriparatide in patients with or without prior antiresorptive treatment: one-year results from the EUROFORS study. Curr Med Res Opin. 2008 Nov;24(11):3117-28. doi: 10.1185/03007990802466595. Epub 2008 Oct 6. PMID 18838053